CLINICAL TRIAL: NCT03233685
Title: Effect of Visual Training on Reaction Time and Timing in Tennis Players
Brief Title: Visual Training and and Reaction Time in Tennis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Matteo Bonato, Matteo Bonato, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Visual Training
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Visuomotor Skills
Keywords: Tennis; Reaction Time; Visual training

STUDY DESIGN:
Intervention Model Description: Randomized control trial.
Who Masked: Participant
Masking Description: The participant will be blind regarding the aim of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Subjects will perform a visual training for 12 weeks
  Interventions: Behavioral: Visual Training
- Control Group (Active Comparator): Subjects will perform the normal training routine for 12 weeks
  Interventions: Behavioral: Normal Training

INTERVENTIONS:
Behavioral: Visual Training — The visual training will be performed 3 times a week for 40 minutes, at the end of warm up and before the technique training. The subjects will be performed a progression of exercise to improve their visual ability, their velocity of interpretation and transformation. The training will be performed with specific panels approved for visual training (S.V.T.A., Torino, Italy).
  Arms: Experimental Group
Behavioral: Normal Training — Normal training routine
  Arms: Control Group

SUMMARY:
Tennis is situational sport in which the result of the game is directly influenced by the interaction with the opponent. In fact, athletes have to respond in a short-time period to change the way of playing by fast analyzing speed, rotation and direction of the tennis ball. Therefore, it is extremely complicated to predict exactly what will happen during games and matches. According to literature goof visual skills, players can receive and process information quickly and can optimize the performance with extreme precision and dexterity. For this reason, visuomotor training aims to improve reaction times, but its efficiency during playing tennis has not yet been investigated. Therefore, the aim of this study is to investigate how this training method could affect the improvement of visuomotor performance in young people between 12 and 18 years old.

DETAILED DESCRIPTION:
Two armed, parallel group, randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years old.
* Playing career of 4 years.

Exclusion Criteria:

* Serious injury in the 6 mouth before the study.
* Subject that already took part to a visual training

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Reaction Time | After 12 weeks of training
  Stroop test

SECONDARY OUTCOMES:
Analysis of tennis skills | After 12 weeks of training
  QLIPP-TM

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bonato, Ph.D., Principal Investigator — University of Milan
Locations (1):
- Università degli Studi di Milano, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No